CLINICAL TRIAL: NCT05176093
Title: A 6-Month Extension Study Following Protocol VMALS-002-2 (A Phase 2a, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety of Engensis in Participants With Amyotrophic Lateral Sclerosis)
Brief Title: A 6-Month Extension Study to Assess the Long-Term Safety of Engensis in Amyotrophic Lateral Sclerosis
Acronym: REViVALS-1B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMALS-002-2b
Record Dates: First submitted 2021-11-05; First posted 2022-01-04 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Engensis (Active Comparator): Active Comparator: Engensis 64 mg Engensis per Treatment Cycle, with each of 3 cycles composed of 2 days of 128 injections each to the right and left target muscles, spaced 2 weeks apart
  Interventions: Biological: Engensis
- Placebo (Placebo Comparator): Placebo Comparator: Placebo 32 mL of Placebo per Treatment Cycle, with each of 3 cycles composed of 2 days of 128 injections each to the right and left target muscles, spaced 2 weeks apart
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Engensis — Lyophilized biologic to be reconstituted containing Engensis
  Arms: Engensis
Other: Placebo — Injectable Liquid
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the long-term safety of intramuscular administration of Engensis in Participants with Amyotrophic Lateral Sclerosis who were previously randomized, received treatment, and completed the Day 180 Visit of Study VMALS-002-2. Safety will be assessed by incidences of treatment-emergent adverse events, treatment emergent serious adverse events, adverse events of special interest, and the clinically significant laboratory values.

DETAILED DESCRIPTION:
VMALS-002-2b was a safety extension study following VMALS-002-2, which was a Phase 2a, double-blind, randomized, placebo-controlled, multicenter study designed to assess the safety of intramuscular administration of Engensis in subjects with Amyotrophic Lateral Sclerosis.Following completion of the Day 180 visit in VMALS-002-2 and signing of written informed consent, subjects were enrolled in this approximately 180-day extension study, with subjects completing combined participation with a Day 365 visit. Assessments to be conducted during this extension study were as follows: vital signs, weight and height, complete physical examination, 12-lead electrocardiogram, a record of all concomitant medications and procedures, clinical laboratory assessments, Revised Amyotrophic Lateral Sclerosis Functional Rating Scale, handheld dynamometry, slow vital capacity, Amyotrophic Lateral Sclerosis Assessment Questionnaire, 40 questions, Patient Global Impression of Change, and Clinical Global Impression of Change. Assessments of treatment-emergent adverse events, treatment-emergent serious adverse events, adverse events of special interest, and clinically significant laboratory values continued from the Day 180 visit of Study VMALS-002-2 through the VMALS-002-2b extension study to Day 365.

ELIGIBILITY:
Inclusion Criteria:

* Participants who complete the Day 180 Visit in VMALS-002-2 are eligible to enroll in this extension study, VMALS-002-2b.

Exclusion Criteria:

- None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-14 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Austin Neuromuscular Center, Austin, Texas, United States
- Hanyang University Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engensis | Placebo
Started | 4 | 4
Completed | 4 | 3
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and Baseline Characteristics (Safety Analysis Population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Engensis | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (16.99) | 52.3 (10.63) | 45.6 (14.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 3 | 2 | 5
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Emergent Adverse Events in More Than 2 Subjects Overall by System Organ Class and Preferred Term
Description: To evaluate the long-term safety of intramuscular injections of Engensis in Participants with Amyotrophic Lateral Sclerosis in more than 2 Participants by System Organ Class and Preferred Term (Safety Analysis Population)
Time Frame: Day 0 to Day 365
Population: Percentages were based on the number of subjects in the Safety Analysis Population by treatment group and overall.
  Subjects were counted once within for each unique Preferred Term.
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 4 | 4
Participants
  Injection site bruising | 3 | 3
  Asthenia | 0 | 2
  Pyrexia | 2 | 1
  Injection site pain | 1 | 1
  Cough | 3 | 1
  Rhinorrhoea | 1 | 1
  Dysphagia | 3 | 2
  Arthralgia | 1 | 1
  Myalgia | 1 | 1
  COVID-19 | 3 | 2
  Headache | 1 | 1

2. Other Pre Specified Outcome: To Evaluate Changes in Muscle Function Following Engensis Injections in Amyotrophic Lateral Sclerosis Participants
Description: Changes from Baseline (Study VMALS 002-2, Day 0) in Revised Amyotrophic Lateral Sclerosis Function Rating TOTAL scores at Day 365 for Engensis compared to Placebo
  There are 12 separate assessments in this neuromuscular assessment covering Bulbar, Fine Motor, Gross Motor and Breathing assessments. Each individual assessment is scored from 0 (worst case) to 4 (best case).
  Total score is calculated as the sum of all 12 assessment subscores. Note that only the Total Score will be reported in the clinical study report due to the small number of subjects.
  The Total Score range is from a minimum of 0 (worst case) to a maximum of 48 (best case).
Time Frame: Day 0 and Day 365
Population: Revised Amyotrophic Lateral Sclerosis Function Rating Total Score and Change from Baseline to Day 365 (Safety Analysis Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 4 | 4
score on a scale
  Baseline - actual value | 39.0 (1.41) | 30.8 (5.62)
  Day 365 / Early Termination - change from baseline | -10.5 (8.23) | -8.7 (9.61)

3. Other Pre Specified Outcome: To Evaluate Muscle Strength Changes Following Engensis Injections in Amyotrophic Lateral Sclerosis Participants
Description: As assessed bilaterally by Hand-Held Dynamometry in muscles in the upper and lower extremities. Muscle Strength as Measured by Handheld Dynamometry (lbs.) and Change from Baseline to Day 365 by Muscle Group (ITT Population)
Time Frame: Day 0 and Day 365
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 4 | 4
Pounds
  Shoulder Flexion-Left - Baseline - Actual | 24.10 (12.572) | 20.08 (11.538)
  Shoulder Flexion-Left - Day 365 - Change from Baseline | -16.13 (12.419) | -8.40 (5.173)
  Shoulder Flexion- Right - Baseline - Actual | 24.645 (11.5448) | 17.850 (12.0423)
  Shoulder Flexion-Right - Day 365 - Change from Baseline | -16.395 (12.8508) | -5.900 (5.1798)
  Elbow Flexion- Left - Baseline - Actual | 29.440 (25.1779) | 14.525 (10.1923)
  Elbow Flexion-Left - Day 365 - Change from Baseline | -20.190 (15.8662) | -5.433 (3.6501)
  Elbow Flexion- Right - Baseline - Actual | 30.53 (26.522) | 13.73 (11.667)
  Elbow Flexion-Right - Day 365 - Change from Baseline | -20.45 (16.083) | -4.1 (1.082)

4. Other Pre Specified Outcome: To Determine Whether Intramuscular Administration of Engensis Has Effects on Respiratory Capacity in Amyotrophic Lateral Sclerosis Participants
Description: Slow vital capacity is a pulmonary function test that quantifies the volume of air that can be slowly exhaled after slow maximum inhalation. It is measured in Liters of air and the percentage of change from baseline is the Percent Predicted Value and Change from Baseline.
  Change from Baseline (Study VMALS 002-2, Day 0) in Slow Vital Capacity on Day 240, Day 300 and Day 365 for Participants with intramuscular administration of Engensis compared to Placebo. Increasing negative Change from Baseline results indicates worsening of respiratory capacity.
Time Frame: Day 0, Day 240, Day 300 and Day 365
Population: Slow Vital Capacity Percent Change from Baseline by Visit (ITT Population)
Measure: Mean (Standard Deviation); unit: percentage of Change from Baseline
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 4 | 4
percentage of Change from Baseline
  Day 240 - Change from Baseline | 0.0 (1.41) | -16.5 (7.78)
  Day 300 - Change from Baseline | -9.3 (11.90) | -7.3 (19.33)
  Day 365/Early Term - Change from Baseline | -17.3 (19.39) | -15.0 (17.52)

5. Other Pre Specified Outcome: To Determine if Intramuscular Engensis Has Effects on Respiratory Function in Amyotrophic Lateral Sclerosis Participants - Tracheostomy
Description: Total participants requiring Tracheostomy procedures that received intramuscular administration of Engensis, compared to total Placebo participants requiring Tracheostomy procedures.
Time Frame: Day 0 to Day 365
Population: Total Tracheostomy procedures for the Safety Analysis Population - Number of Participants - Day 0 to Day 365
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

6. Other Pre Specified Outcome: To Determine if Intramuscular Administration of Engensis Has Positive Effects on Survival in Amyotrophic Lateral Sclerosis Participants - All-Cause Mortality
Description: Total all-cause Mortality for participants that received intramuscular injections of Engensis, compared to total all-cause Mortality for Placebo participants.
  Total participant deaths that received intramuscular administration of Engensis, compared to total Placebo participant deaths.
Time Frame: Day 0 to Day 365
Population: Total all-cause Mortality for participants
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

7. Other Pre Specified Outcome: To Evaluate Quality of Life Improvement Following Engensis Injections in Amyotrophic Lateral Sclerosis Participants Compared to Placebo
Description: The Participant completes the 40 questions in the Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) with 5 categories: Physical Mobility, Activities of Daily Living and Independence, Eating and Drinking, Communication, and Emotional Reactions. Each question has 5 responses to select from: 0-Never (Best Case), 1-Rarely, 2-Sometime, 3-Often, and 4-Always (Worst Case).
  Note for each question there is a Minimum of 0 (Best), to the Maximum 4 (Worst). Decreasing scores indicates improvement of symptoms. The Total Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) scores are per Category as percentages of 100% maximum. Each Category percentage is summed for the Intent-to-treat Population.
  The Change from Baseline was calculated and displayed in the Table. ALSAQ-40 was completed at the pre-dose baseline visit (Day 0), and at the Day 240 and Day 365 visits.
Time Frame: Day 0, Day 240 and Day 365
Population: Percent Change from Baseline (ITT Population) for Engensis and Placebo.
Measure: Mean (Standard Deviation); unit: percentage of Change from Baseline
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 4 | 4
percentage of Change from Baseline
  Day 240 - Physical mobility | 12.5 (2.500) | 3.33 (20.817)
  Day 365/Early Termination - Physical mobility | 13.75 (9.465) | 21.67 (24.664)
  Day 240 - Activities of Daily Living/Independence | 14.17 (11.815) | -.83 (3.819)
  Day 365/Early Termination - Activities of Daily Living/Independence | 21.88 (21.250) | 10.00 (8.660)
  Day 240 - Eating and Drinking | 0 (0) | 11.13 (25.411)
  Day 365/Early Termination - Eating and Drinking | 20.83 (24.994) | 33.33 (28.868)
  Day 240 - Communication | 16.67 (32.036) | 28.57 (6.207)
  Day 365/Early Termination - Communication | 26.80 (33.350) | 32.17 (35.700)
  Day 240 - Emotional Functioning | 3.33 (13.769) | 7.50 (18.875)
  Day 365/Early Termination - Emotional Functioning | 10.00 (24.833) | 12.50 (4.330)

8. Other Pre Specified Outcome: To Evaluate Patient Reported Outcome Improvement Following Engensis Injections in Amyotrophic Lateral Sclerosis Participants Compared to Placebo
Description: The subject's impression of change after treatment was measured with the Patient Global Impression of Change questionnaire through use of the electronic Patient Reported Outcome . This questionnaire measures the subject's perception of how treatment has affected their level of activity, symptoms, emotions, and overall quality of life.
  Each descriptor is ranked on an increasing improvement scale; where 1 = No change (or condition has got worse), 2=Almost the same, hardly any change at all, 3=A little better, but no noticeable change, 4=Somewhat better, but the change has not made any real difference, 5=Moderately better, and a slight but noticeable change, 6=Better, and a definite improvement that has made a real and worthwhile difference, and 7 = A great deal better, and a considerable improvement that as made all the difference.
  The test was self-administered on Days 240 and 365.
Time Frame: Day 240 and Day 365
Population: Patient Global Impression of Change - ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 4 | 4
Participants
  Day 240 - Impression change - or worse: number analyzed (Participants) | 3 | 3
  Day 240 - Impression change - or worse | 2 | 2
  Day 240 - Impression change - Almost the same, hardly any change: number analyzed (Participants) | 3 | 3
  Day 240 - Impression change - Almost the same, hardly any change | 1 | 1
  Day 365/Early termination - Impression change - or worse: number analyzed (Participants) | 4 | 3
  Day 365/Early termination - Impression change - or worse | 4 | 2
  Day 365/Early Termination - Impression change - Almost the same, hardly any change: number analyzed (Participants) | 4 | 3
  Day 365/Early Termination - Impression change - Almost the same, hardly any change | 0 | 1

9. Other Pre Specified Outcome: To Evaluate Clinician Reported Outcome Improvement Following Engensis Injections in Amyotrophic Lateral Sclerosis Participants Compared to Placebo
Description: The Clinical Global Impression of Change is a validated instrument completed by observers as an assessment of Quality of Life. The Clinical Global Impression of Change is an 8-point scale with scores ranging rom Marked Improvement, Moderate Improvement, Minimal Improvement, Slight Improvement, and Unchanged (or Worse), along with an efficacy index with questions in a matrix for therapeutic effect and side effects.The test was completed on Days 240 and 365/ Early Termination.
Time Frame: Day 240 and Day 365
Population: Clinical Global Impression of Change - ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 4 | 4
Participants
  Day 240 - No change: number analyzed (Participants) | 3 | 3
  Day 240 - No change | 2 | 1
  Day 240 - Minimally worse: number analyzed (Participants) | 3 | 3
  Day 240 - Minimally worse | 1 | 1
  Day 240 - Much worse: number analyzed (Participants) | 3 | 3
  Day 240 - Much worse | 0 | 1
  Day 365 / Early Termination - Minimally improved: number analyzed (Participants) | 4 | 3
  Day 365 / Early Termination - Minimally improved | 0 | 1
  Day 365 / Early Termination - No change: number analyzed (Participants) | 4 | 3
  Day 365 / Early Termination - No change | 2 | 0
  Day 365 / Early Termination Minimally worse: number analyzed (Participants) | 4 | 3
  Day 365 / Early Termination Minimally worse | 0 | 1
  Day 365 / Early Termination Much worse: number analyzed (Participants) | 4 | 3
  Day 365 / Early Termination Much worse | 2 | 1

ADVERSE EVENTS:
Time Frame: Day 0 to Day 365, or until participant withdraws informed consent for this extension study, which can be anytime between Day 180 and Day 365.
Description: All study-related Adverse Events will be collected starting after completion of the Informed Consent process at Screening to Day 0/randomization of the VMALS-002-2 study. Treatment-Emergent Adverse Events and Treatment-Emergent Serious Adverse Events will be collected after first injections of VMALS-002-2 study until the time that the Participant withdraws their informed consent for this extension study.
Arm/Group | Engensis | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis (N=4) | Placebo (N=4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral arterialocclusive disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis (N=4) | Placebo (N=4)
Injection site bruising (General disorders) | 3 (6) | 3 (9)
Asthenia (General disorders) | 0 (0) | 2 (4)
Pyrexia (General disorders) | 2 (3) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2)
Injection site pain (General disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyneal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Tachycardia (Vascular disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Bone density descreased (Investigations) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT05176093/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT05176093/SAP_001.pdf